CLINICAL TRIAL: NCT01723046
Title: Active Smart Wearable Orthosis Using Painted EMG Electrodes for Home Based Therapy With Augmentative Feedback
Brief Title: Therapeutic Effects of a New Upper Limb Robot Assisted Therapy Device for Persons After Stroke
Acronym: ARTHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Thomas More Kempen (Other)
Responsible Party: Principal Investigator, Lore Van de Perre, Study principal investigator, Thomas More Kempen
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IWT120278
Record Dates: First submitted 2012-10-30; First posted 2012-11-07 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Stroke
Keywords: Upper extremity; Rehabilitation; Robot assisted therapy; Robotics; Devices; Orthosis; clinical outcome
MeSH Terms: conditions — Stroke | interventions — Exoskeleton Device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training with the device (Experimental): Training with new upper limb robot assisted therapy device
  Interventions: Device: Training with new upper limb robot assisted therapy device
- Control group (No Intervention): The control group is treated with conventional therapy.

INTERVENTIONS:
Device: Training with new upper limb robot assisted therapy device — During 8 weeks, 3 times a week, 1 hour therapy sessions with the device
  Other Names: active orthosis; exoskeleton
  Arms: Training with the device

SUMMARY:
The purpose of this pilot study is to investigate the clinical effects of a new upper limb robot assisted therapy device that is linked to a virtual therapy environment in patients with stroke.

DETAILED DESCRIPTION:
The number of physically weak individuals is increasing, resulting in a higher burden on health care and health care workers. The use of robot assisted therapy (RAT) might partly solve this problem. Rehabilitation progress highly depends on training intensity and training duration, favouring the use of RAT.

In this pilot study, the clinical effects of using a new upper arm RAT device for upper arm rehabilitation in patients with stroke is investigated. Myo-electrical signals will serve as input for the device, assisting the user in flexion and extension of the elbow. The device is coupled to a virtual environments, creating a stimulating therapy environment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stroke, more than three months post onset
* No or moderate spasticity in the upper limb (maximum score of 3 on Modified Ashworth Scale)
* Observable voluntary muscle activity in biceps and triceps muscle of the affected upper limb (minimal score of 1 on the Medical research council score)
* Able to sit on a chair with adequate trunk stability
* Able to follow verbal instructions
* Able to communicate verbal information to the researchers

Exclusion Criteria:

* Patients who are medically unstable
* Cognitive disorders impeding the intervention
* Visual disorders impeding the intervention
* Subluxation of the shoulder joint
* Pusher syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer test upper limb section | Change from baseline Fugl-Meyer test upper limb section at 8 weeks and 12 weeks
  Stroke specific, performance based impairment index. Applied to determine disease severity and describe motor recovery.
Medical research council score | Change from baseline Medical research council score at 8 weeks and 12 weeks
  Muscle strength assessment
Active range of motion of the elbow joint | Change from baseline active range of motion of the elbow joint at 8 weeks and 12 weeks
  The maximum range of motion to flexion and extension of the elbow joint that the person can achieve independently
Passive range of motion of the elbow joint | Change from baseline passive range of motion of the elbow joint at 8 weeks and 12 weeks
  The maximum range of motion to flexion and extension of the elbow joint of the test person that can be achieved by the assessor.
Modified Ashworth Scale | Change from baseline Modified Ashworth Scale at 8 weeks and 12 weeks
  Spasticity measurement

SECONDARY OUTCOMES:
ABILHAND questionnaire | Change from baseline ABILHAND questionnaire score at 8 weeks and 12 weeks
  Questionnaire-based assessment of manual ability
Functional independence measure | Change from baseline Functional independence measure score at 8 weeks and 12 weeks
  Assessment of physical and cognitive disability, focusing on the burden of care.
Stroke impact scale | Change from baseline Stroke impact scale score at 8 weeks and 12 weeks
  Questionnaire evaluating how stroke has impacted the person's health and life.
Intrinsic motivation inventory | Change from baseline Intrinsic motivation inventory score at 8 weeks and 12 weeks
  Multidimensional measurement device intended to assess participants' subjective experience related to a target activity in laboratory experiments.

CONTACTS AND LOCATIONS:
Overall Officials: Lore Van de Perre, MSc, Principal Investigator — Thomas More Kempen
Locations (1):
- Thomas More Kempen, Geel, Antwepen, Belgium